CLINICAL TRIAL: NCT06067126
Title: PrepareD: Examining Post-Delivery Maternal-offspring Obesity and Metabolic Risk After a Prepregnancy Weight-loss Intervention
Brief Title: Post-delivery Maternal-offspring Obesity and Metabolic Risk After a Prepregnancy Weight-loss Intervention
Acronym: PrepareD
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: 5R01DK125348 (NIH); 5R01DK125348 (NIH)
Record Dates: First submitted 2023-08-13; First posted 2023-10-04 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Overweight; Obese; Metabolic Disorders; Postpartum
Keywords: Wellness/Behavior Change
MeSH Terms: conditions — Overweight; Obesity; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of PrepareD is to examine whether the prepregnancy weight-loss intervention administered during the Prepare trial [NCT02346162] has an influence in the postnatal period. PrepareD is a cohort study (no intervention) that will address new specific aims through one in-person visit with mothers and children, dietary recalls, actigraphy, and the use of medical record weights. The goal is to collect data when the child is 3 years old. However, due to the COVID-19 pandemic, the investigators expanded the data collection window in order to collect data up to when the child is 5 years old. The investigators hypothesize that intervening on women before pregnancy is the key to breaking the multigenerational cycle of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Mother must be a Prepare [NCT02346162] participant who has experienced a viable pregnancy during the Prepare trial
* Child must be the first viable offspring born to a Prepare participant after consent into the Prepare study

Exclusion Criteria: None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants for PrepareD will be recruited from the pool of women who consented to participate in the Prepare trial [NCT02346162]. The investigators expect to re-enroll around 180 Prepare mother-offspring pairs in the PrepareD study.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Child body mass index (BMI) from birth up to 5 years of age | Birth up to 5 years of age
  All child weights, lengths (before age 2), and heights (after age 2) recorded in the electronic medical record (EMR) between delivery and up to 5 years of age will be collected. Child weight and height between 3 years 0 months of age up until 5 years of age will be measured at an in-person research visit. Weight in kilograms (kg) and height in meters (m) will be combined to report BMI in kg/m^2.
Mother postpartum weight retention (PPWR) in pounds at 5 weeks and 1 year postpartum | 5 weeks and 1 year after delivery
  All weights recorded for the mother in the EMR between delivery and up to 5 weeks and 1 year postpartum will be collected. PPWR at 5 weeks and 1 year after delivery will be obtained by subtracting mother's 5-week postpartum weight (in lbs) and 1-year postpartum weight (in lbs) from mother's weight (in lbs) at delivery, respectively.

SECONDARY OUTCOMES:
Healthy Eating Index (HEI) score for mother and child | At study visit, when child is 3-4 years of age
  Mother and child dietary data will be collected via dietary recalls following the study visit in order to calculate HEI total and component scores for mother and child.
Daily activity level for mother and child | At study visit, when child is 3-4 years of age
  Mother and child activity level will be collected via actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Erin S LeBlanc, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Any information from this study presented in reports or publications will not identify any individual.